CLINICAL TRIAL: NCT06691399
Title: Routine Oral Care Versus Chlorhexidine Oral Care on Incidence of Nosocomial Pneumonia and Oral Health Among Critically Ill Non-intubated Patients With COPD
Brief Title: Role of Oral Care in Prevention of Nosocomial Pneumonia Among COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant Professor of Chest Diseases, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SOD2024
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Nosocomial Pneumonia; COPD Exacerbation
Keywords: COPD; Oral care; Nosocomial pneumonia; Chlorhexidine
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pulmonary Disease, Chronic Obstructive | interventions — Dental Care Team

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine oral care (Group 1) (Placebo Comparator): Group (1) will receive routine oral care twice daily with gauze for cleansing and tooth brushing
  Interventions: Other: Oral care
- Chlorhexidine oral care (Active Comparator): Group (1) will receive routine oral care twice daily with gauze for cleansing and tooth brushing plus oral care with chlorohexidine solution (concentration 1.2%)
  Interventions: Other: Oral care

INTERVENTIONS:
Other: Oral care — Oral care done twice daily with chlorhexidine oral care solution (concentration 1.2%)

SUMMARY:
Poor dental hygiene has been linked to respiratory pathogen colonization in ICU patients. Therefore, respiratory pathogens tend to colonize dental plaque and oral mucosa in these populations. Therefore, strategies to eliminate respiratory pathogens from the oral cavity may improve oral hygiene and decrease the development of nosocomial pneumonia.

DETAILED DESCRIPTION:
Infection is a common problem and a major cause of morbidity and mortality for patients in intensive care units (ICUs). Pneumonia is the most common site of infection according to an international study of the prevalence and outcomes of infection in ICUs, which included 13,796 patients. Nosocomial pneumonia (NP) is among the leading causes of mortality in patients in the ICU. Notably, the incidence of nosocomial pneumonia is increasing, and the number of infection-related deaths that follow is also increasing. Thus, preventing nosocomial pneumonia is a cost reducing and life-saving health care practice, especial in ICUs.

Nosocomial pneumonia (NP) was defined as an infection of the lower respiratory tract that does not exist at the time of admission and does not have an incubation period of infection but occurs 48 hours after admission. The most important cause for the development of nosocomial pneumonia is the oral environment. The oral cavity of ICU patients is an important reservoir for bacteria and provides a habitat for microorganisms that can lead to nosocomial pneumonia. Patients in ICUs acquire pneumonia by aspirating oral bacteria that have been colonized in the oral cavity into the lower respiratory tract. Due to advanced age, limited mobility, illness, and cognitive dysfunction, patients in ICUs often have difficulty maintaining oral hygiene by themselves.

Poor dental hygiene has been linked to respiratory pathogen colonization in ICU patients. Therefore, respiratory pathogens tend to colonize dental plaque and oral mucosa in these populations. Therefore, strategies to eliminate respiratory pathogens from the oral cavity may improve oral hygiene and decrease the development of nosocomial pneumonia. The aim of the present study is to assess value of preventive strategy using chlorhexidine for oral care among non-intubated COPD patients admitted to ICU upon incidence of nosocomial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as COPD
* admitted to ICU with acute exacerbation
* need for noninvasive ventilatory support including noninvasive ventilation anf high flow nasal cannula

Exclusion Criteria:

* patients refusing to participate
* End stage organ failure (Heart Failure, Liver cell failure and/or Renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of nosocomial pneumonia | 1 month
  Incidence of nosocomial pneumonia diagnosed via clinical features and confirmed with either chest ultrasonography or chest radiography

CONTACTS AND LOCATIONS:
Overall Officials: Waleed MD Gamal Elddin Khaleel, Ass. Prof., Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Vilela MC, Ferreira GZ, Santos PS, Rezende NP. Oral care and nosocomial pneumonia: a systematic review. Einstein (Sao Paulo). 2015 Apr-Jun;13(2):290-6. doi: 10.1590/S1679-45082015RW2980. Epub 2015 May 1. PMID 25946053